CLINICAL TRIAL: NCT04563793
Title: Postmarket Outcomes Study for Evaluation of the Superion™ Spacer
Acronym: PRESS2
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: A4086
Record Dates: First submitted 2020-09-17; First posted 2020-09-24 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-09

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Superion™ IDS: All patients to receive IDS for the treatment of their moderate Lumbar Spinal Stenosis Symptoms.
  Interventions: Device: Superion™ IDS

INTERVENTIONS:
Device: Superion™ IDS — All patients to receive IDS for the treatment of moderate Lumbar Spinal Stenosis symptoms.

SUMMARY:
To compile real-world outcomes of the Superion™ IDS in routine clinical practice.

DETAILED DESCRIPTION:
The purpose of this outcomes study is to compile real-world outcomes for the commercially approved Indirect Decompression Systems (IDS) in routine clinical practice when used according to the applicable Instructions for Use.

ELIGIBILITY:
Key Inclusion Criteria:

* Scheduled to receive or previously received a commercially approved Boston Scientific Indirect Decompression Systems, per local Instructions for Use (IFU)
* Signed a valid, IRB approved informed consent form

Key Exclusion Criteria:

* Meets any contraindication in BSC Indirect Decompression Systems local IFU

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with moderate Lumbar Spinal Stenosis
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, Study Director — Boston Scientific Corporation
Locations (23):
- United States (23):
  - Pain Medicine Associates, Fountain Valley, California
  - California Orthopedics & Spine, Larkspur, California
  - Relieve Pain Center, Inc., San Diego, California
  - Source Healthcare, Santa Monica, California
  - Pacific Research Institute, Santa Rosa, California
  - IPM Medical Group Inc, Walnut Creek, California
  - Holy Cross Hospital Inc., Fort Lauderdale, Florida
  - Louis J. Raso, MD, PA, Jupiter, Florida
  - Florida Pain Institute, Merritt Island, Florida
  - Southwest Florida Pain Center, Port Charlotte, Florida
  - Georgia Pain and Spine Care, Inc., Newnan, Georgia
  - Centurion Spine and Pain Centers, Waycross, Georgia
  - North Idaho Day Surgery LLC, Post Falls, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - KC Pain Centers, Lee's Summit, Missouri
  - Comprehensive and Interventional Pain Management LLP, Henderson, Nevada
  - Premier Pain Center, Shrewsbury, New Jersey
  - University Clinical Research Center, Somerset, New Jersey
  - The Toledo Clinic, Toledo, Ohio
  - Center for Interventional Pain and Spine, Bryn Mawr, Pennsylvania
  - Advanced Spine Pain Solution, Laredo, Texas
  - Precision Spine Care, Tyler, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Superion™ IDS: All patients to receive IDS for the treatment of their moderate Lumbar Spinal Stenosis Symptoms.
  Superion™ IDS: All patients to receive IDS for the treatment of moderate Lumbar Spinal Stenosis symptoms.
  Patients include previously implanted subjects and newly enrolled subjects up to 3 years post-procedure.
Period: Overall Study
Arm/Group | Superion™ IDS
Started | 129
Completed | 23
Not Completed | 106

BASELINE CHARACTERISTICS:
Population: All subjects who completed the baseline information. Two subjects were consented but did not complete the baseline information.
Arm/Group | Superion™ IDS
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: American Indian or Alaska native | 2
  Race/Ethnicity: Black, of African heritage | 5
  Race/Ethnicity: Caucasian | 104
  Race/Ethnicity: Hispanic or Latino | 8
  Race/Ethnicity: Other | 2
  Race/Ethnicity: Not disclosed | 6
Region of Enrollment [Number; unit: participants]
  United States | 127
Low Back pain/symptoms [Count of Participants; unit: Participants] — Percentage of patients with low back pain/symptoms
  Participants | 124

OUTCOME MEASURES:

1. Primary Outcome: Low Back Pain Responder Rate
Description: Proportion of subjects with an improvement of 20 mm during the last 7 days for low back pain at 6 months, 1 year, 2 years, and 3 years post-procedure compared with Baseline (VAS)
Time Frame: Up to 3 years post-procedure
Population: Intent-to-Treat (ITT) Population: Patients who receive treatment with the Superion® Indirect Decompression System (IDS).
  Patients include previously implanted subjects and newly enrolled subjects up to 3 years post-procedure. Data for patients previously implanted includes data which was collected retrospectively.
Measure: Count of Participants; unit: Participants
Groups:
- Superion™ IDS 6-Month Follow-up: All patients to receive IDS for the treatment of their moderate Lumbar Spinal Stenosis Symptoms and completed 6-Month Visit.
- Superion™ IDS 1-Year Follow-up: All patients to receive IDS for the treatment of their moderate Lumbar Spinal Stenosis Symptoms and completed 1-Year Visit.
- Superion™ IDS 2-Year Follow-up: All patients to receive IDS for the treatment of their moderate Lumbar Spinal Stenosis Symptoms and completed 2-Year Visit.
- Superion™ IDS 3-Year Follow-up: All patients to receive IDS for the treatment of their moderate Lumbar Spinal Stenosis Symptoms and completed 3-Year Visit.
Arm/Group | Superion™ IDS 6-Month Follow-up | Superion™ IDS 1-Year Follow-up | Superion™ IDS 2-Year Follow-up | Superion™ IDS 3-Year Follow-up
Number analyzed (Participants) | 30 | 11 | 8 | 7
Participants | 17 | 3 | 1 | 2

2. Primary Outcome: Left Leg Pain Responder Rate
Description: Proportion of subjects with an improvement of 20 mm during the last 7 days for left leg pain at 6 months, 1 year, 2 years, and 3 years post-procedure compared with Baseline (VAS)
Time Frame: Up to 3 years post-procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Superion™ IDS 6-Month Follow-up | Superion™ IDS 1-Year Follow-up | Superion™ IDS 2-Year Follow-up | Superion™ IDS 3-Year Follow-up
Number analyzed (Participants) | 23 | 9 | 4 | 5
Participants | 15 | 7 | 2 | 0

3. Primary Outcome: Right Leg Pain Responder Rate
Description: Proportion of subjects with an improvement of 20 mm during last 7 days for left leg pain at 6 months, 1 year, 2 years, and 3 years post-procedure compared with Baseline (VAS)
Time Frame: Up to 3 years post-procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Superion™ IDS 6-Month Follow-up | Superion™ IDS 1-Year Follow-up | Superion™ IDS 2-Year Follow-up | Superion™ IDS 3-Year Follow-up
Number analyzed (Participants) | 25 | 10 | 7 | 6
Participants | 18 | 6 | 3 | 0

4. Other Pre Specified Outcome: Percent Low Back Pain Relief
Description: Percent Low Back Pain Relief at 6 months, 1 year, 2 years and 3 years post-procedure compared with Baseline (PPR).
  PPR is a questionnaire assessing how much of the subject's low back pain has been relieved by treatment. Pain relief is expressed as a percentage from 0 - 100%.
Time Frame: Up to 3 years post-procedure
Population: No patients completed the percent pain relief at 2 and 3-Year Follow-up Visits. Intent-to-Treat (ITT) Population: Patients who receive treatment with the Superion® Indirect Decompression System (IDS).
  Patients include previously implanted subjects and newly enrolled subjects up to 3 years post-procedure. Data for patients previously implanted includes data which was collected retrospectively.
Measure: Mean (Standard Deviation); unit: percentage of low back pain relief
Arm/Group | Superion™ IDS 6-Month Follow-up | Superion™ IDS 1-Year Follow-up
Number analyzed (Participants) | 33 | 10
percentage of low back pain relief | 46.7 (37.4) | 58.3 (42.2)

5. Other Pre Specified Outcome: Quality of Life (QoL)
Description: Percent of change from Baseline index score to the Follow-up timepoints index score using EQ-5D-5L.
  EuroQol Five Dimensions Five Level questionnaire (EQ-5D-5L) is comprised of a descriptive system and a visual analog scale (VAS). The descriptive system measures quality of life along five dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with five levels for each dimension from which subjects are asked to select one. VAS is used to record the subject's self-rated health on a 20cm vertical line with endpoints labeled 'the best health you can imagine' and 'the worst health you can imagine'. To calculate the Index Value, responses are converted into a single score using a specific algorithm. Score ranges from 0.000 (representing death) to 1.000 (representing perfect health). The algorithm is based on public preferences, reflecting how different health states are valued by the general public.
Time Frame: Up to 3 years post-procedure
Population: No patients completed EQ5D-5L at 2 and 3 year visits. Intent-to-Treat (ITT) Population: Patients who receive treatment with the Superion® Indirect Decompression System (IDS).
  Patients include previously implanted subjects and newly enrolled subjects up to 3 years post-procedure. Data for patients previously implanted includes data which was collected retrospectively.
Measure: Mean (Standard Deviation); unit: percent change of score on a scale
Arm/Group | Superion™ IDS 6-Month Follow-up | Superion™ IDS 1-Year Follow-up
Number analyzed (Participants) | 34 | 12
percent change of score on a scale | 65.6 (89.2) | 47.8 (44.6)

ADVERSE EVENTS:
Time Frame: From the time a subject sign the PRESS 2 Study Informed Consent through 3-year visit or study withdrawal. Patients include previously implanted subjects and newly enrolled subjects up to 3 years post-procedure. Data for patients previously implanted includes retrospective data however adverse events were monitored/assess from the time a subject signed the PRESS 2 Study Informed Consent through study completion.
Description: Other (Not including Serious) Adverse Events definition differs from clinicaltrials.gov results Data Element definition - Per the study protocol, only device hardware and/or procedure related adverse events were monitored/assessed. Other, non-serious adverse events not related to the device hardware and/or procedure were not collected or assessed in this study.
  All Serious Adverse Events and All-Cause Mortality were monitored/assessed per the clinicaltrials.gov definition.
Arm/Group | Superion™ IDS
All-Cause Mortality (participants affected / at risk) | 0/129
Serious Adverse Events (participants affected / at risk) | 12/129
Other Adverse Events (participants affected / at risk) | 3/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Superion™ IDS (N=129)
Spinal Fracture (Injury, poisoning and procedural complications) | 1
Acute coronary syndrome (Cardiac disorders) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Spinal operation (Surgical and medical procedures) | 1 (1)
Deep Vein thrombosis (Vascular disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Superion™ IDS (N=129)
Purulent discharge (Infections and infestations) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT04563793/Prot_SAP_000.pdf